CLINICAL TRIAL: NCT03334864
Title: Observational Cohort Study of Advanced Non-small Cell Lung Cancer (CAPTRA-LUNG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-1410
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-11

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: Advanced non-small cell lung cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- I Retrospective cohort: Diagnosis of advanced non-small cell lung cancer from 2012-2016
- II Prospective cohort: Advanced non-small cell lung cancer with driver gene mutations
- III Prospective cohort: Non-small cell lung cancer in immuno-therapy;
- IV Prospective cohort: Non-small cell lung cancer with wild-type driver gene or unknown driver gene status;
- V Prospective cohort: Advanced non-small lung cancer with wild-type gene treated with anti-Vascular Endothelial Growth Factor (VEGF) drug.

SUMMARY:
Investigators propose to establish and maintain a cohort of patients with advanced non-small cell lung cancer, and to assess the treatment pattern, host genetic, and clinical factors which influence the prognosis and survival, as well as the interaction among these factors on disease diagnosis and treatment, short and long-term outcomes.

Study type: Observational (Patient Registry)

Study design: Observational Model: Cohort

Time Perspective: Prospective and retrospective

ELIGIBILITY:
Inclusion Criteria:

* Cohort I: diagnosis of advanced non-small cell lung cancer from 2012-2016;
* Cohort II: documented positive driver gene mutations; and diagnosis of advanced non-small cell lung cancer;
* Cohort III: diagnosis of advanced non-small cell lung cancer and in immune-therapy;
* Cohort IV: diagnosis of advanced non-small cell lung cancer, and with wild-type driver gene or unknown driver gene status;
* Cohort V: treated with anti-VEGF drug in first line, diagnosis of advanced non-squamous and non-small cell lung cancer in 6 months before recruit;
* Age>18 years;
* Provision of written informed consent.

Exclusion Criteria:

* not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5000 advanced NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years
  OS was calculated from the diagnosis of advanced non-small cell lung cancer to death from any reasons

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Y, Zhang L, Fang J, Wang Z, Li J, Li L, Ai B, Nie L, Mu X, Liang L, Zhang S, Zhang Y, Song Y, Song X, Wang Y, Xin T, Jin B, Wang X, Ding C, Wang M. Establishment of a prospective multicenter cohort for advanced non-small cell lung cancer in China (CAPTRA-Lung study). Thorac Cancer. 2018 Dec;9(12):1795-1800. doi: 10.1111/1759-7714.12865. Epub 2018 Sep 27. PMID 30264504